CLINICAL TRIAL: NCT02890966
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of SHR4640 in Healthy Subjects
Brief Title: Multiple Dose Study of SHR4640 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-102
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Gout; Hyperuricemia
Keywords: SHR4640 pharmacokinetics pharmacodynamics
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 1mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: placebo
- Cohort 2 (Experimental): 2.5mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: placebo
- Cohort 3 (Experimental): 5mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: placebo
- Cohort 4 (Experimental): 10mg SHR4640 or placebo
  Interventions: Drug: SHR4640; Drug: placebo

INTERVENTIONS:
Drug: SHR4640 — Day1~Day7:oral administration
Drug: placebo — Day1~Day7:oral administration

SUMMARY:
The objective of the study is to assess the tolerance, pharmacokinetic and pharmacodynamic properties of multiple dose adminstration of SHR4640 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55, male;
2. Body weight≥50, BMI:19-25kg/m2;

3.4 mg/dL≤Screening serum urate level≤7 mg/dL;

4.Medically stable based on physical examination, laboratory results, vital sign measurements, 12-lead electrocardiogram, abdomen B-ultrasound and Chest X-ray examination at screening.

Exclusion Criteria:

1. Serum creatinine>upper limits of normal(ULN);
2. Alanine aminotransferase and/or Aspartate aminotransferase>2×ULN, total bilirubin>1.5×ULN, glutamyltransferase>3×ULN;
3. History of hyperuricemia or gout;
4. History or suspicion of kidney stones;
5. Positive results for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, syphilis antibody test.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | Clinical significant changes from baseline up to Day 10

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax)(of single dose and at stable status) | Up to Day 10
Area under the plasma concentration versus time curve(AUC)(of single dose and at stable status) | Up to Day 10
Half-time(T1/2)(of single dose and at stable status) | Up to Day 10
Time to the peak plasma concentration(Tmax)(of single dose and at stable status) | Up to Day 10
Changes in serum uric acid concentration from baseline | Up to Day 10
Changes in urinary uric acid excretion from baseline | Up to Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- The South West Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided